CLINICAL TRIAL: NCT01883999
Title: Evaluation of the GORE® EXCLUDER® Iliac Branch Endoprosthesis for the Treatment of Common Iliac Artery Aneurysms or Aorto-iliac Aneurysms
Brief Title: Evaluation of the GORE® EXCLUDER® Iliac Branch Endoprosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBE 12-04
Record Dates: First submitted 2013-06-18; First posted 2013-06-21 (Estimated); Results first posted 2016-08-03 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Common Iliac Artery Aneurysms; Aorto-iliac Aneurysms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GORE® EXCLUDER® Iliac Branch Endoprosthesis (Experimental): GORE® EXCLUDER® Iliac Branch Endoprosthesis
  Interventions: Device: GORE® EXCLUDER® Iliac Branch Endoprosthesis

INTERVENTIONS:
Device: GORE® EXCLUDER® Iliac Branch Endoprosthesis

SUMMARY:
The Iliac Branch Endoprosthesis (IBE) 12-04 study will be a prospective, nonrandomized, multicenter, single-arm evaluation designed to assess the safety and efficacy of the IBE Device in subjects with common iliac artery aneurysms (CIAA) or aorto-iliac aneurysms (AIA).

ELIGIBILITY:
Inclusion Criteria:

1. Common iliac aneurysm with or without concomitant abdominal aortic aneurysm
2. Adequate native anatomy to receive the EXCLUDER® and Iliac Branch Endoprostheses
3. An Informed Consent Form signed by Subject or legally authorized representative
4. Male or infertile female
5. Able to comply with protocol requirements including following-up
6. Life expectancy > 2 years
7. Age > 21 years
8. Surgical candidate

Exclusion Criteria:

1. Mycotic or ruptured aneurysm
2. Known concomitant thoracic aortic aneurysm which requires intervention
3. American Society of Anesthesiologists (ASA) Physical Status classification system class V (moribund patient not expected to live 24 hours with or without operation)
4. Renal insufficiency defined or patient undergoing dialysis
5. New York Heart Association (NYHA) Functional Classification class IV
6. Dissected, heavily calcified, or heavily thrombosed landing zone(s)
7. Tortuous or stenotic iliac and/or femoral arteries
8. Participating in another investigational device or drug study within 1 year of treatment
9. Systemic infection which may increase the risk of endovascular graft infection
10. Known degenerative connective tissue disease, e.g., Marfan or Ehler-Danlos Syndrome
11. Planned concomitant surgical procedure or major surgery within 30 days of treatment date
12. Known history of drug abuse
13. Known sensitivities or allergies to the device materials

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2021-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darren Schneider, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Schneider DB, Matsumura JS, Lee JT, Peterson BG, Chaer RA, Oderich GS. Five-year outcomes from a prospective, multicenter study of endovascular repair of iliac artery aneurysms using an iliac branch device. J Vasc Surg. 2023 Jan;77(1):122-128. doi: 10.1016/j.jvs.2022.07.006. Epub 2022 Jul 13. PMID 35842202
- [Derived] Schneider DB, Milner R, Heyligers JMM, Chakfe N, Matsumura J. Outcomes of the GORE Iliac Branch Endoprosthesis in clinical trial and real-world registry settings. J Vasc Surg. 2019 Feb;69(2):367-377.e1. doi: 10.1016/j.jvs.2018.05.200. Epub 2018 Jul 29. PMID 30064841

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GORE® EXCLUDER® Iliac Branch Endoprosthesis
Started | 64
Completed | 61
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | GORE® EXCLUDER® Iliac Branch Endoprosthesis
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 63
Region of Enrollment [Number; unit: participants]
  United States | 64

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Composite of the Following: Death, Stroke, Myocardial Infarction, Bowel Ischemia, Paraplegia, Respiratory Failure, Renal Failure, Conversion to Open Surgical Repair
Description: Freedom from composite of the following: Death, Stroke, Myocardial Infarction, Bowel Ischemia, Paraplegia, Respiratory Failure, Renal Failure, Conversion to open surgical repair.
Time Frame: 30 days post-treatment
Population: Subjects initiating IBE procedure and meeting inclusion/exclusion criteria
Measure: Number; unit: participants
Arm/Group | GORE® EXCLUDER® Iliac Branch Endoprosthesis
Number analyzed (Participants) | 62
participants | 62

2. Primary Outcome: Freedom From: Reintervention on Iliac Branch Component (IBC) or Internal Iliac Component (IIC) Due to Type I/III Endoleak or to Re-establish Patency Due to 60% Occlusion or Greater, or Complete Loss of Blood Flow in Leg of IBC or IIC
Description: Freedom from all of the following:
  * Reintervention on Iliac Branch Component (IBC) or Internal Iliac Component (IIC) due to Type I/III endoleak as determined by Clinical Events Committee (CEC).
  * Complete loss of blood flow in leg of IBC or IIC as assessed by Core Laboratory
  * Reintervention on IBC or IIC to re-establish patency due to 60% occlusion or greater as determined by CEC.
Time Frame: Through 6 month follow-up visit
Population: Subjects having IBC and IIC components implanted and meeting inclusion/exclusion criteria
Measure: Number; unit: participants
Arm/Group | GORE® EXCLUDER® Iliac Branch Endoprosthesis
Number analyzed (Participants) | 61
participants | 58

3. Secondary Outcome: Freedom From New Onset Buttock Claudication Arising From the Side of the Body Treated With the Iliac Branch Component (IBC) and Internal Iliac Component (IIC)
Description: Freedom from new onset buttock claudication arising from the side of the body treated with the Iliac Branch Component (IBC) and Internal Iliac Component (IIC).
Time Frame: Through 6 month follow-up visit
Population: Subjects having IBC and IIC components implanted and meeting inclusion/exclusion criteria
Measure: Number; unit: participants
Arm/Group | GORE® EXCLUDER® Iliac Branch Endoprosthesis
Number analyzed (Participants) | 61
participants | 61

ADVERSE EVENTS:
Time Frame: 6 months or more of follow-up
Description: All follow-up at time of endpoint calculation for subjects undergoing IBE Device procedure (6 months post-treatment and later if available)
Arm/Group | GORE® EXCLUDER® Iliac Branch Endoprosthesis
Serious Adverse Events (participants affected / at risk) | 25/63
Other Adverse Events (participants affected / at risk) | 53/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GORE® EXCLUDER® Iliac Branch Endoprosthesis (N=63)
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Stent-graft endoleak (General disorders) | 1
Thrombosis in device (General disorders) | 1
Contrast media allergy (Immune system disorders) | 1
Incision site infection (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Hip fracture (Injury, poisoning and procedural complications) | 1
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Aortic dissection (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Peripheral artery aneurysm (Vascular disorders) | 1
Peripheral artery dissection (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GORE® EXCLUDER® Iliac Branch Endoprosthesis (N=63)
Stent-graft endoleak (General disorders) | 27
Urinary tract infection (Infections and infestations) | 4
Incision site pain (Injury, poisoning and procedural complications) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 7
Urinary retention (Renal and urinary disorders) | 5
Intermittent claudication (Vascular disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other